CLINICAL TRIAL: NCT06712394
Title: Interspace Between the Popliteal Artery and Capsule of the Posterior Knee-
Brief Title: Knee Osteoarthritis and IPACK
Acronym: IPACK
Status: Not yet recruiting | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Other Study IDs: isik eman ipack
Record Dates: First submitted 2024-09-03; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IPACK: IPACK block involves ultrasound-guided local anesthetic infiltration of the space between the popliteal artery and the posterior knee joint capsule.
  Interventions: Procedure: IPACK

INTERVENTIONS:
Procedure: IPACK — The IPACK block involves infiltration of the space between the popliteal artery and the posterior knee joint capsule with 20 ml of 0.25% local anesthetic (bupivacain) under ultrasound guidance.

SUMMARY:
Interspace between the Popliteal Artery and Capsule of the posterior Knee (IPACK) block involves ultrasound-guided local anesthetic infiltration of the space between the popliteal artery and the posterior knee joint capsule.

The purpose of the study; To investigate the effectiveness of this block applied to knee osteoarthritis in clinical practice.

In this study, patients who underwent IPACK block by the practitioner; Demographic data, medications used, block success, block characteristics and block-related complications will be recorded observationally. Before and after the block procedure, patients' pain was measured with the Numeric Rating Scale (NRS) at 1st and 3rd months, their disability levels were measured with The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire and Short Form-12 (Short Form). Quality of life will be measured with the -SF-12) survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from grade 3 and 4 knee osteoarthritis

Exclusion Criteria:

* Patients who have had previous knee surgery
* Patients who have had any knee injection in the last 3 months
* Malignancy
* Inflammatory disease
* Infectious disease (local or general)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50-90 who underwent IPACK block treatment due to Knee OA
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 1st and 3rd month after the procedure
  The Numeric Rating Scale (NRS) is a frequently used tool for assessing and monitoring the severity of pain. The pain scale measures on an 11-point rating system, where 0 indicates the absence of pain and 10 represents the most severe pain one can imagine. Patients are requested to assess their pain on a scale ranging from 0 to 10. The physician obtained from measurements at each visit by directly questioning the patient.
Functional status | 1st and 3rd month after the procedure
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of knee osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain, stiffness, and physical function. The questionnaire evaluates activities of daily living and functional mobility. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Quality of life assessment | 1st and 3rd month after the procedure
  The assessment of quality of life was conducted using the SF-12, a questionnaire specifically designed to measure health-related quality of life. The SF-12 consists of twelve items that evaluate eight different health domains, providing an evaluation of both physical and mental well-being. The SF-12 provides two summary scores: the mental component score (MCS-12) and the physical component score (PCS-12). A decrease in the questionnaire score indicates progression of disability. The questionnaire's validity and reliability were ensured, and the Turkish version of the questionnaire was filled out by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rıdvan Isık, Study Chair — sakarya training and research hospital, pain clinic